CLINICAL TRIAL: NCT00102167
Title: A Double-Blind, Randomized, Placebo-Controlled, Parallel-Group, Multicenter Study of MK0928 in Healthy Adult Volunteers Participating in a 4-Hour Phase Advance Model of Transient Insomnia
Brief Title: Study of MK0928 in Healthy Adult Volunteers in a Model of Insomnia (0928-006)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Executive Vice President, Clinical and Quantitative Sciences, Merck Sharp & Dohme Corp
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0928-006; MK0928-006; 2004_092
Record Dates: First submitted 2005-01-21; First posted 2005-01-24 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — gaboxadol

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: gaboxadol — Duration of Treatment -1 day
  Other Names: MK0928

SUMMARY:
A study to evaluate the safety and effectiveness of Study of MK0928 in Healthy Adult Volunteers in a Model of Insomnia for insomnia (a sleep disorder).

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults who are between the ages of 18 and 64

Exclusion Criteria:

* Adults who are diagnosed with insomnia

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 663 (Actual)
Dates: Start 2005-02; Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Amount of time spent awake and time to fall asleep during one night | one night

SECONDARY OUTCOMES:
Amount of deep sleep during one night. | one night
Patient-reported sleep quality and awakenings during 1 night. | one night

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Walsh JK, Mayleben D, Guico-Pabia C, Vandormael K, Martinez R, Deacon S. Efficacy of the selective extrasynaptic GABA A agonist, gaboxadol, in a model of transient insomnia: a randomized, controlled clinical trial. Sleep Med. 2008 May;9(4):393-402. doi: 10.1016/j.sleep.2007.06.006. Epub 2007 Aug 30. PMID 17765013
- [Derived] Ma J, Dijk DJ, Svetnik V, Tymofyeyev Y, Ray S, Walsh JK, Deacon S. EEG power spectra response to a 4-h phase advance and gaboxadol treatment in 822 men and women. J Clin Sleep Med. 2011 Oct 15;7(5):493-501A. doi: 10.5664/JCSM.1316. PMID 22003345